CLINICAL TRIAL: NCT05004779
Title: Regenerative Effects of Human Stem Cell Media After Laser Therapy in Hypertrophic Scar Caused by Burns
Brief Title: Regenerative Effects of Human Stem Cell Media After Laser Therapy in Hypertrophic Scar
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hangang Sacred Heart Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HangangSHH-13
Record Dates: First submitted 2021-07-29; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-07

CONDITIONS: Stem Cell Media; Hypertrophic Scar; Regeneration
Keywords: stem cell media; non ablative laser; hypertrophic scar; burns; regeneration
MeSH Terms: conditions — Cicatrix, Hypertrophic; Burns

STUDY DESIGN:
Intervention Model Description: After laser treatment on hypertrophic scars, human stem cell conditioned media was applied to one side and physiological saline was applied to the other side.
Who Masked: Participant
Masking Description: After laser treatment on hypertrophic scars, human stem cell media was applied to one side and physiological saline was applied to the other side.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- human stem cell media apply lesion (Experimental): human media apply after non ablative laser treatment
  Interventions: Procedure: human stem cell conditioned media was applied after non-ablative laser therapy
- control condition lesion (Sham Comparator): normal saline apply after non ablative laser treatment
  Interventions: Procedure: normal saline was applied after non ablative laser therapy

INTERVENTIONS:
Procedure: human stem cell conditioned media was applied after non-ablative laser therapy — After laser treatment on hypertrophic scars, human stem cell media was applied to one side
  Arms: human stem cell media apply lesion
Procedure: normal saline was applied after non ablative laser therapy — physiological saline was applied to the other side.
  Arms: control condition lesion

SUMMARY:
The purpose of this study was to determine the effect of combined treatment using nonablative laser and human stem cell media (HSCM) on the regeneration of hypertrophic scars that occurred after burns.

DETAILED DESCRIPTION:
The purpose of this study was to determine the effect of combined treatment using nonablative laser and human stem cell media (HSCM) on the regeneration of hypertrophic scars that occurred after burns. Nonablative laser treatment was performed on 30 patients with hypertrophic scars on both sides of the same part of the body. Immediately after the laser treatment, the hypertrophic scars of right side to which HSCM was applied and the left side with the same body position were defined as a control scar, and normal saline was applied. Over the next 6 days, HSCM and moisturizer were applied on the scars of right side, and only moisturizer was applied on the control scar of left side. Laser treatment was performed three times on the hypertrophic scar at 4 weeks intervals. The skin test on hypertrophic scar was evaluated before laser treatment and re-evaluated on the 7the day after the 3rd laser treatment. The thickness was measured with a ultrasonic wave equipment (128 BW1 Medison, Korea). Mexameter® (MX18, Courage-Khazaka Electronics GmbH, Germany) was used to measure melanin levels and the severity of erythema. The higher values indicating a darker and redder skin. Transepidermal water loss (TEWL) was measured with a Tewameter® (Courage-Khazaka Electronic GmbH, Germany), which is used for evaluating water evaporation. Sebum in the scars was measured with the Sebumeter® (Courage-Khazaka Electronic GmbH, Germany). The measurement is based on the principle of grease-spot photometry using a cassette with its special tape. A microprocessor calculates the result, which is shown on the display in μg/cm2. Elasticity was measured using Cutometer SEM 580® (Courage-Khazaka Electronic GmbH, Cologne, Germany), which applies negative pressure (450 mbar) on the skin. The numeric values (mm) of the skin's distortion is presented as the elasticity (Table 1). Two seconds of negative pressure of 450 mbar is followed by 2 s of recess, and this consists of a complete cycle. Three measurement cycles were conducted, and the average values were obtained. To evaluate the effect of HSCM, investigators compared the skin test results (thickness, melanin, erythema, TEWL, sebum, and skin elasticity levels) between the right side and control side, from baseline measures immediately before the laser treatment and measures on the 7the day after the 3rd laser treatment. Outcome measurements and data analyses were performed by a trained and blinded outcome assessor who was not involved in the intervention. Possible complications (pain, ecchymosis, skin abrasion, and swelling) were observed.

ELIGIBILITY:
Inclusion Criteria:

* partial or full-thickness burns that healed spontaneously or required skin grafting
* with hypertrophic scars on the right and left sides of the same body part

Exclusion Criteria:

* Patients with open wounds or infection on the burn scars
* those taking steroids for the scars
* with allergies to topical anesthetic cream
* those who were pregnant
* undergoing any other medical treatment or condition affecting wound healing (e.g., diabetes)

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-10 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-04-20 (Estimated)

PRIMARY OUTCOMES:
scar thickness (cm) | baseline
  The thickness was measured with a ultrasonic wave equipment
change from baseline scar thickness at 3 months (cm) | after 3 months intervention
  the change of scar thickness was measured with a ultrasonic wave equipment

SECONDARY OUTCOMES:
melanin levels (arbitraty units; AU) | baseline
  the higher values indicating a darker
change from baseline melanin level at 3 months (arbitraty units; AU) | after 3 months intervention
  the higher values indicating a darker
erythema level (arbitraty units; AU) | baseline
  the higher values indicating a redder skin
change from baseline erythema level at 3 months (arbitraty units; AU) | after 3 months intervention
  the higher values indicating a redder skin
transepidermal water loss (g/h/m2) | baseline
  the higher the number, the more dry the skin is.
change from baseline transepidermal water loss at 3 months (g/h/m2) | after 3 months intervention
  the higher the number, the more dry the skin is.
Sebum level (μg sebum/cm2) | baseline
  A microprocessor calculates the result, which is shown on the display in μg/cm2. The higher the number, the more oily the skin is.
change from baseline sebum level at 3 months (μg sebum/cm2) | after 3 months intervention
  A microprocessor calculates the result, which is shown on the display in μg/cm2. The higher the number, the more oily the skin is.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Onur Erol O, Agaoglu G, Jawad MA. Combined Non-Ablative Laser and Microfat Grafting for Burn Scar Treatment. Aesthet Surg J. 2019 Mar 14;39(4):NP55-NP67. doi: 10.1093/asj/sjy291. PMID 30403775
- [Result] Jayaraman P, Nathan P, Vasanthan P, Musa S, Govindasamy V. Stem cells conditioned medium: a new approach to skin wound healing management. Cell Biol Int. 2013 Oct;37(10):1122-8. doi: 10.1002/cbin.10138. Epub 2013 Jun 24. PMID 23716460
- [Result] Park IS. Enhancement of Wound Healing by Conditioned Medium of Adipose-Derived Stromal Cell with Photobiomodulation in Skin Wound. Int J Stem Cells. 2021 May 30;14(2):212-220. doi: 10.15283/ijsc20175. PMID 33632992